CLINICAL TRIAL: NCT00258596
Title: Sirolimus-Eluting Stents for Chronic Total Coronary Occlusions: A Randomized Comparison of Bare Metal Stent Implantation With Sirolimus-Eluting Stent Implantation for the Treatment of Chronic Total Coronary Occlusions (PRISON II)
Brief Title: Sirolimus-Eluting Stents for Chronic Total Coronary Occlusions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: R&D Cardiologie (Other)
Collaborators: Cordis US Corp. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RDC-2002-01-PRISON II
Record Dates: First submitted 2005-11-23; First posted 2005-11-24 (Estimated); Last update posted 2007-03-06 (Estimated); Status verified 2007-01

CONDITIONS: Coronary Artery Disease; Coronary Disease; Coronary Stenosis
Keywords: drug-eluting stent; chronic total occlusion; sirolimus-eluting stent; zotarolimus-eluting stent; QCA
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Coronary Stenosis

INTERVENTIONS:
Device: sirolimus-eluting stent

SUMMARY:
Primary intracoronary stent placement after successfully crossing chronic total occlusions (CTO) decreases the high restenosis rate at long-term follow-up compared with conventional balloon angioplasty. Several studies have shown the efficacy of sirolimus-eluting stents in selected groups of patients. Whether sirolimus-eluting stents are superior to bare metal stents in CTO is unknown. In this prospective randomized trial, bare metal stent implantation will be compared with sirolimus-eluting stent implantation for the treatment of chronic total coronary occlusions. A total of 200 patients will be followed up for 6, 12, and 24 months with angiographic follow-up at 6 months. Quantitative coronary analysis will be performed by an independent core laboratory. The primary end point is the binary angiographic restenosis and reocclusion rate at 6 month follow-up.

DETAILED DESCRIPTION:
Since data from the 2 landmark studies, the BENESTENT and STRESS studies, showed that coronary stenting significantly decreases restenosis as compared with conventional balloon angioplasty, this treatment modality has shown to be superior in an increasing number of indications. Percutaneous coronary intervention of chronic total occlusions (CTO), however, is still limited by high restenosis rates. Although coronary stenting using bare metal stents significantly decreases restenosis in CTO, restenosis rates still reach 32% to 55%.

In 200 patients with CTO randomized in the PRISON I study, we demonstrated a restenosis rate of 22% after bare metal stent implantation as compared with 33% after conventional balloon angioplasty. During the past few years, sirolimus (rapamycin), a cytostatic macrocyclic lactone with anti-inflammatory and antiproliferative properties, delivered from a polymer-encapsulated stent was shown to almost eliminate the risk of restenosis in selected groups of patients.

In this prospective, randomized, single-blind trial we enrolled 200 patients with chronic total occlusions: 100 were randomly assigned to receive bare metal BxVelocity™ stents, and 100 to receive sirolimus-eluting Cypher™ stents. The primary endpoint was angiographic binary restenosis rate at six months follow-up. Secondary endpoints were a composite of major adverse cardiac events, target vessel failure, in-stent and in-segment minimal lumen diameter, percentage diameter stenosis, and late luminal loss at six months follow-up. Clinical long-term follow-up will performed up till 24 months

ELIGIBILITY:
Inclusion Criteria:

* Estimated duration of the chronic total coronary occlusion of at least two weeks
* Evidence of ischemia related to the target vessel (signs of ischemia during an abnormal exercise test, defined as ST depression of at least 1.0 mm that is horizontal or down-sloping or up-sloping ST depression of at least 2.0 mm or signs of ischemia found during nuclear imaging with exercise, dobutamine or adenosine).

Exclusion Criteria:

* The lesion could not be crossed
* The use of heparin, aspirin and clopidogrel was prohibited
* Severe renal failure (creatinine>250µmol/L)
* Patients were unwilling or unable to complete follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2003-01; Study Completion 2006-09

PRIMARY OUTCOMES:
The binary restenosis rate (defined as restenosis >50% on follow-up angiography) at six-month angiography

SECONDARY OUTCOMES:
A composite of: Major adverse cardiac events (death, myocardial infarction, and ischemia driven target lesion revascularization)
Target vessel failure (defined as a composite of death from cardiac causes, myocardial infarction, and ischemia-driven target-vessel revascularization) at 6 month
In-stent and in-segment minimal lumen diameter
Percentage in-stent and in-segment diameter stenosis
In-stent and in-segment late luminal loss at six months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Maarten J. Suttorp, MD, PhD, Principal Investigator — St. Antonius Hospital
Locations (2):
- Netherlands (2):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - St Antonius Hospital, Nieuwegein

REFERENCES:
- [Background] Rahel BM, Suttorp MJ, Laarman GJ, Kiemeneij F, Bal ET, Rensing BJ, Ernst SM, ten Berg JM, Kelder JC, Plokker HW. Primary stenting of occluded native coronary arteries: final results of the Primary Stenting of Occluded Native Coronary Arteries (PRISON) study. Am Heart J. 2004 May;147(5):e22. doi: 10.1016/j.ahj.2003.11.023. PMID 15131557
- [Background] Suttorp MJ, Mast EG, Plokker HW, Kelder JC, Ernst SM, Bal ET. Primary coronary stenting after successful balloon angioplasty of chronic total occlusions: a single-center experience. Am Heart J. 1998 Feb;135(2 Pt 1):318-22. doi: 10.1016/s0002-8703(98)70099-7. PMID 9489982
- [Background] Serruys PW, de Jaegere P, Kiemeneij F, Macaya C, Rutsch W, Heyndrickx G, Emanuelsson H, Marco J, Legrand V, Materne P, et al. A comparison of balloon-expandable-stent implantation with balloon angioplasty in patients with coronary artery disease. Benestent Study Group. N Engl J Med. 1994 Aug 25;331(8):489-95. doi: 10.1056/NEJM199408253310801. PMID 8041413
- [Background] Fischman DL, Leon MB, Baim DS, Schatz RA, Savage MP, Penn I, Detre K, Veltri L, Ricci D, Nobuyoshi M, et al. A randomized comparison of coronary-stent placement and balloon angioplasty in the treatment of coronary artery disease. Stent Restenosis Study Investigators. N Engl J Med. 1994 Aug 25;331(8):496-501. doi: 10.1056/NEJM199408253310802. PMID 8041414
- [Background] Rensing BJ, Vos J, Smits PC, Foley DP, van den Brand MJ, van der Giessen WJ, de Feijter PJ, Serruys PW. Coronary restenosis elimination with a sirolimus eluting stent: first European human experience with 6-month angiographic and intravascular ultrasonic follow-up. Eur Heart J. 2001 Nov;22(22):2125-30. doi: 10.1053/euhj.2001.2892. PMID 11686669
- [Background] Moses JW, Leon MB, Popma JJ, Fitzgerald PJ, Holmes DR, O'Shaughnessy C, Caputo RP, Kereiakes DJ, Williams DO, Teirstein PS, Jaeger JL, Kuntz RE; SIRIUS Investigators. Sirolimus-eluting stents versus standard stents in patients with stenosis in a native coronary artery. N Engl J Med. 2003 Oct 2;349(14):1315-23. doi: 10.1056/NEJMoa035071. PMID 14523139
- [Background] Sirnes PA, Golf S, Myreng Y, Molstad P, Emanuelsson H, Albertsson P, Brekke M, Mangschau A, Endresen K, Kjekshus J. Stenting in Chronic Coronary Occlusion (SICCO): a randomized, controlled trial of adding stent implantation after successful angioplasty. J Am Coll Cardiol. 1996 Nov 15;28(6):1444-51. doi: 10.1016/s0735-1097(96)00349-x. PMID 8917256
- [Background] Rahel BM, Laarman GJ, Suttorp MJ; PRISON II study investigators. Primary stenting of occluded native coronary arteries II--rationale and design of the PRISON II study: a randomized comparison of bare metal stent implantation with sirolimus-eluting stent implantation for the treatment of chronic total coronary occlusions. Am Heart J. 2005 Mar;149(3):e1-3. doi: 10.1016/j.ahj.2004.10.027. PMID 15864219
- [Derived] Rahel BM, Laarman GJ, Kelder JC, Ten Berg JM, Suttorp MJ. Three-year clinical outcome after primary stenting of totally occluded native coronary arteries: a randomized comparison of bare-metal stent implantation with sirolimus-eluting stent implantation for the treatment of total coronary occlusions (Primary Stenting of Totally Occluded Native Coronary Arteries [PRISON] II study). Am Heart J. 2009 Jan;157(1):149-55. doi: 10.1016/j.ahj.2008.08.025. Epub 2008 Nov 6. PMID 19081412